CLINICAL TRIAL: NCT05384626
Title: A Phase 1/2 Study of the Selective Anaplastic Lymphoma Kinase (ALK) Inhibitor NVL-655 in Patients With Advanced NSCLC and Other Solid Tumors (ALKOVE-1)
Brief Title: A Study of Neladalkib (NVL-655) in Patients With Advanced NSCLC and Other Solid Tumors Harboring ALK Rearrangement or Activating ALK Mutation (ALKOVE-1)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nuvalent Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NVL-655-01
Expanded Access: NCT06834074 (Available)
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Locally Advanced Solid Tumor; Metastatic Solid Tumor
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Phase 1 dose escalation (Experimental): Neladalkib (NVL-655) oral daily dosing
  Interventions: Drug: Neladalkib (NVL-655)
- Cohort 2a (Experimental): Patients with locally advanced or metastatic NSCLC harboring an ALK rearrangement who have received 1 prior 2nd-generation ALK TKI (ceritinib, alectinib, or brigatinib). Up to 2 prior lines of chemotherapy and/or immunotherapy are allowed.
  Interventions: Drug: Neladalkib (NVL-655)
- Cohort 2b (Experimental): Patients with locally advanced or metastatic NSCLC harboring an ALK rearrangement, who have received 2-3 prior ALK TKIs (crizotinib, ceritinib, alectinib, brigatinib, or lorlatinib). Up to 2 prior lines of chemotherapy and/or immunotherapy are allowed.
  Interventions: Drug: Neladalkib (NVL-655)
- Cohort 2c (Experimental): Patients with locally advanced or metastatic NSCLC harboring an ALK rearrangement, who have received lorlatinib as the only prior ALK TKI therapy. Up to one prior line of chemotherapy and/or immunotherapy received prior to lorlatinib is allowed.
  Interventions: Drug: Neladalkib (NVL-655)
- Cohort 2d (Experimental): Patients with locally advanced or metastatic NSCLC harboring an ALK rearrangement, who are naïve to ALK TKI therapy. Up to one prior line of chemotherapy and/or immunotherapy is allowed.
  Interventions: Drug: Neladalkib (NVL-655)
- Cohort 2e (Experimental): Patients with locally advanced or metastatic NSCLC harboring an ALK rearrangement, not eligible for other Phase 2 cohorts.
  Interventions: Drug: Neladalkib (NVL-655)
- Cohort 2f (Experimental): Patients with other solid tumors harboring an ALK rearrangement or activating ALK mutation, who have received ≥1 prior systemic anticancer therapy, or for whom no satisfactory standard therapy exists.
  Interventions: Drug: Neladalkib (NVL-655)

INTERVENTIONS:
Drug: Neladalkib (NVL-655) — Oral Tablet of Neladalkib (NVL-655)

SUMMARY:
Phase 1/2, dose escalation and expansion study designed to evaluate the safety and tolerability of neladalkib (NVL-655), determine the recommended phase 2 dose (RP2D), and evaluate the antitumor activity in patients with advanced ALK- positive (ALK+) NSCLC and other solid tumors.

Phase 1 will evaluate the overall safety and tolerability of neladalkib and will determine the RP2D and, if applicable, the maximum tolerated dose (MTD) of neladalkib in patients with advanced ALK+ solid tumors.

Phase 2 will determine the objective response rate (ORR) as assessed by Blinded Independent Central Review (BICR) of neladalkib at the RP2D. Secondary objectives will include the duration of response (DOR), time to response (TTR), progression-free survival (PFS), overall survival (OS), and clinical benefit rate (CBR) of neladalkib in patients with advanced ALK-positive NSCLC and other solid tumors.

DETAILED DESCRIPTION:
In Phase 2, study patients will be enrolled into 6 distinct cohorts:

* Cohort 2a: Patients with locally advanced or metastatic NSCLC harboring an ALK rearrangement who have received 1 prior 2nd-generation ALK TKI (ceritinib, alectinib, or brigatinib). Up to 2 prior lines of chemotherapy and/or immunotherapy are allowed.
* Cohort 2b: Patients with locally advanced or metastatic NSCLC harboring an ALK rearrangement, who have received 2-3 prior ALK TKIs (crizotinib, ceritinib, alectinib, brigatinib, or lorlatinib). Up to 2 prior lines of chemotherapy and/or immunotherapy are allowed.
* Cohort 2c: Patients with locally advanced or metastatic NSCLC harboring an ALK rearrangement, who have received lorlatinib as the only prior ALK TKI therapy. Up to one prior line of chemotherapy and/or immunotherapy received prior to lorlatinib is allowed.
* Cohort 2d: Patients with locally advanced or metastatic NSCLC harboring an ALK rearrangement, who are naïve to ALK TKI therapy. Up to one prior line of chemotherapy and/or immunotherapy is allowed.
* Cohort 2e: Patients with locally advanced or metastatic NSCLC harboring an ALK rearrangement, not eligible for other Phase 2 cohorts.
* Cohort 2f: Patients with other solid tumors harboring an ALK rearrangement or activating ALK mutation, who have received ≥1 prior systemic anticancer therapy, or for whom no satisfactory standard therapy exists.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, Phase 2 Cohort 2f only: Age ≥12 years and weighing >40 kg.
2. Phase 1: Histologically or cytologically confirmed locally advanced or metastatic solid tumor with a documented ALK rearrangement or activating ALK mutation.
3. Phase 2

   1. Phase 2 Cohorts except 2f: Histologically or cytologically confirmed locally advanced or metastatic NSCLC with a documented ALK rearrangement
   2. Phase 2 Cohort 2f: Histologically or cytologically confirmed locally advanced or metastatic solid tumor with a documented ALK rearrangement or activating ALK mutation detected by certified assay.
4. Phase 1: Must have evaluable disease (target or nontarget) according to RECIST 1.1 Phase 2: Must have measurable disease according to RECIST 1.1
5. Adequate organ function and bone marrow reserve

Exclusion criteria:

1. Patient's cancer has a known oncogenic driver alteration other than ALK.
2. Known allergy/hypersensitivity to excipients of NVL-655.
3. Major surgery within 4 weeks of the study entry
4. Ongoing or anticancer therapy
5. Actively receiving systemic treatment or direct medical intervention on another therapeutic clinical study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 840 (Estimated)
Dates: Start 2022-06-09 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLTs) (Phase 1) | Within the first 21 days of the first neladalkib (NVL-655) dose
  Define the dose limiting toxicities (DLTs)
Recommended Phase 2 Dose (RP2D) (Phase 1) | Within 21 days of last patient dosed during escalation
  To determine the RP2D
Objective Response Rate (ORR) (Phase 2) | 2-3 years after first patient dosed.
  To determine ORR as assessed by BICR
Number of participants with treatment-emergent adverse events, as assessed by CTCAE, V5.0 (Phase 1) | Approximately 3 years
  Incidence and severity of treatment-emergent adverse events (TEAEs)

SECONDARY OUTCOMES:
Maximum plasma concentration, (Cmax) of neladalkib (NVL-655) | Pre-dose and up to 24 hours post-dose
  To determine the maximum plasma concentration (Cmax) of neladalkib (NVL-655)
Plasma concentration at the end of the dosing interval (Ctau) of neladalkib (NVL-655) | Pre-dose and up to 24 hours post-dose
  To determine the plasma concentration at the end of the dosing interval (Ctau) of neladalkib (NVL-655)
Average plasma concentration (Cavg) of neladalkib (NVL-655) | Pre-dose and up to 24 hours post-dose
  To determine the average plasma concentration (Cavg) of neladalkib (NVL-655)
Time of maximum concentration (Tmax) of neladalkib (NVL-655) | Pre-dose and up to 24 hours post-dose
  To determine the time of maximum concentration (Tmax) of neladalkib (NVL-655)
Area under the curve at the end of the dosing interval (AUCtau) of neladalkib (NVL-655) | Pre-dose and up to 24 hours post-dose
  To determine the area under the curve at the end of the dosing interval (AUCtau) of neladalkib (NVL-655)
Area under the curve from time 0 to 24 (AUC0-24) of neladalkib (NVL-655) | Pre-dose and up to 24 hours post-dose
  To determine the area under the curve from time 0 to 24 (AUC0-24) of neladalkib (NVL-655)
Area under the curve from time 0 to infinity (AUCinf) of neladalkib (NVL-655) | Pre-dose and up to 24 hours post-dose
  To determine the area under the curve from time 0 to infinity (AUCinf) of neladalkib (NVL-655)
Oral clearance (CL/F) of neladalkib (NVL-655) | Pre-dose and up to 24 hours post-dose
  To determine the oral clearance (CL/F) of neladalkib (NVL-655)
Volume of distribution (Vz/F) of neladalkib (NVL-655) | Pre-dose and up to 24 hours post-dose
  To determine the volume of distribution (Vz/F) of neladalkib (NVL-655)
Half-life (t1/2) of neladalkib (NVL-655) | Pre-dose and up to 24 hours post-dose
  To determine the half-life (t1/2) of neladalkib (NVL-655)
Objective response rate (ORR) (Phase 1) | 2-3 years after first patient dosed
  Determine ORR as assessed by Investigator
Duration of response (DOR) | 2-3 years after first patient dosed
  Determine DOR of neladalkib (NVL-655) until radiographic disease progression or death
Clinical benefit rate (CBR) | 2-3 years after first patient dosed
  Determine CBR of neladalkib (NVL-655)
Time to response | Approximately 3 years
  Determine time to response of neladalkib (NVL-655)
Progression-free survival (PFS) | 2-3 years after first patient dosed
  Determine PFS of neladalkib (NVL-655) until radiographic disease progression or death
Overall survival (OS) (Phase 2) | Approximately 3 years
  Determine OS
Number of participants with treatment-emergent adverse events, as assessed by CTCAE, V5.0 (Phase 2) | Approximately 3 years
  Incidence and severity of treatment-emergent adverse events (TEAEs)
Quality of life assessment | 2-3 years after first patient dosed
  Measure the quality of life in patients with cancer and/or lung cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Viola Zhu, MD, PHD, Study Director — Nuvalent Inc.
Locations (74):
- United States (21):
  - University of California Irvine Medical Center, Orange, California
  - University of California, Davis Comprehensive Cancer Center, Sacramento, California
  - Stanford Cancer Institute, Stanford, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - University of Miami; Sylvester Cancer Center, Miami, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - John Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Cancer Institute, Detroit, Michigan
  - Washington University School of Medicine Siteman Cancer Center, St Louis, Missouri
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - OSU Brain & Spine Hospital, Columbus, Ohio
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Australia (3):
  - Royal North Shore Hospital, Sydney, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Belgium (2):
  - Universitair Ziekenhuis Antwerpen (UZA), Antwerp
  - Universitaire Ziekenhuizen Leuven Campus Gastthuisberg, Leuven
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer Center, Vancouver, British Columbia
  - The Ottawa Hospital Cancer Center, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
- France (4):
  - Centre Leon Berard, Lyon
  - Chu De Nantes, Nantes
  - Institut Claudius Regaud, Toulouse
  - Institute Gustave Roussy, Villejuif
- Germany (4):
  - Universitatsklinikum Koln - University Hospital Cologne, Cologne
  - Universitätsklinikum Frankfurt, Frankfurt
  - LungenClinic Grosshansdorf GmbH, Großhansdorf
  - Universkitatsklinikum Heidelberg - University Hospital Heidelberg, Heidelberg
- Italy (7):
  - Azienda Ospedaliera Universitaria Ospedali Riuniti Umberto, Ancona
  - IRCCS Istituto Tumori "G. Paolo II", Bari
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Instituto Europeo di Oncologia, Milan
  - Instituto Oncologico Veneto, Padua
  - Ospedale Santa Maria delle Croci, Ravenna
  - Regina Elena Institute for Cancer Research, Rome
- Japan (7):
  - Kanagawa Cancer Center, Kanagawa
  - Okayama University Hospital, Okayama
  - Kindai University Hospital, Osaka
  - Shizuoka Cancer Center, Shizuoka
  - National Cancer Center Hospital, Tokyo
  - Cancer Institute Hospital of JFCR, Tokyo
  - Wakayama Medical University Hospital, Wakayama
- Netherlands (2):
  - The Netherlands Cancer Institute, Amsterdam
  - University Medical Center Groningen (UMCG), Groningen
- Singapore (2):
  - National University Hospital, Singapore, Singapore
  - National Cancer Centre Singapore, Singapore, Singapore
- South Korea (4):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
- Spain (5):
  - Complejo Hospitalario Universitario de A Coruna, A Coruña
  - UOMI Cancer Center, Barcelona
  - Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Switzerland (2):
  - Istituto Oncologico Svizzera Italiana, Bellinzona
  - Luzerner Kantonsspital, Lucerne
- Taiwan (3):
  - Chung-Shan Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- United Kingdom (4):
  - Royal Marsden Hospital, Sutton, Surrey
  - Edinburgh Cancer Centre, Edinburgh
  - The Royal Marsden - Chelsea, London
  - The Christie NHS Foundation Trust, Manchester